CLINICAL TRIAL: NCT01928212
Title: Retinal Nerve Fiber Layer Thickness Changes in Parkinson Disease: A Meta-analysis
Status: Completed | Type: Observational
Sponsor: Yifan Feng (Other)
Collaborators: Wenzhou Medical University (Other)
Responsible Party: Sponsor-Investigator, Yifan Feng, Eye Hospital, Wenzhou Medical College, China, Wenzhou Medical University
Organization: Wenzhou Medical University (Other)
Other Study IDs: FYF20130820
Record Dates: First submitted 2013-08-20; First posted 2013-08-23 (Estimated); Last update posted 2014-07-18 (Estimated); Status verified 2014-07

CONDITIONS: Parkinson Disease
Keywords: retinal nerve fiber layer thickness; optical coherence tomography; Parkinson disease
MeSH Terms: conditions — Parkinson Disease | interventions — Tomography, Optical Coherence

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective

GROUPS / COHORTS (2):
- healthy control: Sex- and agematched healthy subjects
  Interventions: Device: Optical coherence tomography
- Parkinson group: Patients with Parkinson's disease
  Interventions: Device: Optical coherence tomography

INTERVENTIONS:
Device: Optical coherence tomography

SUMMARY:
Optical coherence tomography (OCT) is a non-invasive retinal imaging technology that can provide high-resolution cross-sectional images of the peripapillary retinal nerve fiber layer (RNFL) and measure its thickness. A reduction of the RNFL thickness has been detected in several neurodegenerative diseases, such as multiple sclerosis, CADASIL and Alzheimer's disease. Different studies have reported RNFL changes also in Parkinson's disease (PD),a common neurodegenerative disease characterized by motor dysfunctions, originally described by James Parkinson in 1817. PD is characterized by selective dopaminergic neuronal cells loss, which may correlate with RNFL thinning. Previous studies on this subject, however, reported contradicting results. Some investigations reported reductions of the RNFL thickness while others did not. In the present study, in order to determine whether RNFL thickness is reduced in PD patients, we performed a meta-analysis and systematically evaluated RNFL thickness measurements with OCT in a series of PD patients and in the healthy control groups.

ELIGIBILITY:
Inclusion Criteria:

1. case-control studies;
2. patients with PD were compared with healthy controls;
3. all subjects underwent RNFL thickness measurement by OCT;
4. studies should provide the data of peripapillary RNFL thickness;
5. sample size ≥10 in each group.

Exclusion Criteria:

1. authors did not make RNFL measurements;
2. study without healthy control group;
3. the outcome values can not be used for meta-analysis;
4. duplicated articles.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: PD patients and healthy subjects were included and underwent OCT examinations
Sampling Method: Probability Sample
Enrollment: 500 (Actual)
Dates: Start 2013-08; Primary Completion 2014-01 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
Retinal Nerve Fiber Layer Thickness | Baseline
  Retinal nerve fiber layer thickness included average thickness (360° measurement), temporal quadrant thickness (316-45°), superior quadrant thickness (46-135°), nasal quadrant thickness (136-225°) and inferior quadrant thickness (226-315°)was measured by OCT.

CONTACTS AND LOCATIONS:
Overall Officials: Yifan Feng, PhD, Principal Investigator — Wenzhou Medical University
Locations (1):
- Wenzhou Medical College, Wenzhou, Zhejiang, China

REFERENCES:
- [Derived] Yu JG, Feng YF, Xiang Y, Huang JH, Savini G, Parisi V, Yang WJ, Fu XA. Retinal nerve fiber layer thickness changes in Parkinson disease: a meta-analysis. PLoS One. 2014 Jan 21;9(1):e85718. doi: 10.1371/journal.pone.0085718. eCollection 2014. PMID 24465663